CLINICAL TRIAL: NCT07386730
Title: A Double Blind, Randomized Trial Investigating the Safety, Feasibility, and Mechanisms of Psychedelics in Healthy Older Adults With Low Well-being as Moderated by Biomarkers for Preclinical Alzheimer's Disease
Brief Title: A Study of Psychedelics in Healthy Older Adults With Low Well-being
Acronym: OAD1
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jennifer Mitchell (Other)
Responsible Party: Sponsor-Investigator, Jennifer Mitchell, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25-45261; A146672 (Other Grant/Funding Number: Brain & Behavior Research Foundation)
Record Dates: First submitted 2026-01-20; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Anhedonia in Healthy Volunteers; Older Adults (50-90 Years)
Keywords: Psilocybin; Dextromethorphan; older adults; well-being; EEG; MRI; neuroinflammation; Alzheimer's disease plasma markers; wearables
MeSH Terms: conditions — Neuroinflammatory Diseases | interventions — Psilocybin; Pharmaceutical Preparations; Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A low-to-moderate dose of Psilocybin (5-10 mg) (Experimental): A single low-to-moderate dose of Psilocybin (5-10 mg)
  Interventions: Drug: Psilocybin (drug)
- A moderate-to-high dose of Psilocybin (25-30 mg) (Experimental): A single moderate-to-high dose of Psilocybin (25-30 mg)
  Interventions: Drug: Psilocybin (drug)
- A low-to-moderate dose of Dextromethorphan (30-60 mg) (Experimental): A single low-to-moderate dose of Dextromethorphan (30-60 mg)
  Interventions: Drug: Dextromethorphan (DXM)
- A moderate-to-high dose of Dextromethorphan (80-90 mg) (Experimental): A single moderate-to-high dose of Dextromethorphan (80-90 mg)
  Interventions: Drug: Dextromethorphan (DXM)

INTERVENTIONS:
Drug: Psilocybin (drug) — Participants will receive either Psilocybin or Dextromethorphan in this clinical trial
  Arms: A low-to-moderate dose of Psilocybin (5-10 mg); A moderate-to-high dose of Psilocybin (25-30 mg)
Drug: Dextromethorphan (DXM) — Participants will receive either Psilocybin or Dextromethorphan in this clinical trial
  Arms: A low-to-moderate dose of Dextromethorphan (30-60 mg); A moderate-to-high dose of Dextromethorphan (80-90 mg)

SUMMARY:
This study is being conducted to understand changes in brain activity following administration of two different drugs (Psilocybin and Dextromethorphan) in older adults with low well-being.

The main questions it aims to answer are, does psilocybin:

1. Acutely increase complexity of EEG activity in older adults with low well-being, as modulated by the presence of biomarkers of Alzheimer's disease (AD) pathology.
2. Longitudinally decrease plasma markers of neuroinflammation, as modulated by the presence of biomarkers of AD pathology.
3. Explore longitudinal changes in autonomic physiology via wearable recording devices as well as longitudinal structural and functional brain changes measured in the MRI

Participants will be in the study for up to 3 months, which will include 3 to 4 in person visits and 3 to 4 remote visits. Most visits will be between 1 to 3 hours, but the dosing visit will last a minimum of 8 hours and could be as long as 12 hours. During the dosing visit, all participants will receive a single dose of the study drugs and dosages listed below.

Researchers will compare participants who receive the following drug options:

* A low-to-moderate dose of Psilocybin (5-10 mg)
* A moderate-to-high dose of Psilocybin (25-30 mg)
* A low-to-moderate dose of Dextromethorphan (30-60 mg)
* A moderate-to-high dose of Dextromethorphan (80-90 mg)

ELIGIBILITY:
The eligibility criteria are deliberately incomplete to preserve the scientific integrity of the study.

Inclusion Criteria:

* Are between 50-85 years inclusive at time of consent signing
* Have below-average well-being, defined by the World Health Organization Well-Being Index (WHO-5)
* Have no cognitive impairments, indicated by a Mini-Mental State Examination (MMSE) score >24
* Have an identified willing contact person with at least weekly contact with the participant to be able to provide meaningful information about the participant's daily function and able to pick up the study participant at the end of the Dosing Visit
* Participants assigned female sex at birth must be non-lactating, and post-menopausal, defined as a period of over 12 months since the last menstrual period, or otherwise physically unable to become pregnant
* Participants assigned male sex at birth must 1) refrain from sperm donation for 3 months after the Dosing Visit, and 2) if engaging in sexual activities that may result in pregnancy, must use a condom, plus their partner of childbearing potential must use a second, highly effective form of contraception for 3 months after the Dosing Visit
* Be proficient in English
* Are able and willing to provide consent as assessed by comprehension questions in informed consent process
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Ability to swallow oral medications (capsules)

Exclusion Criteria:

General:

* Have a known allergic or severe reaction to Psilocybin, Dextromethorphan, or any of the non-active components of the IMP capsules
* Insufficient ability to report on symptoms to make a valid assessment on any required instrument
* Have a condition or presence of clinical feature which, in the opinion of the investigators might interfere with or prevent appropriate study participation or interfere with data interpretation

MRI Exclusions:

* Any implanted object or device that poses a safety risk or could interfere with MRI scanning (e.g. aneurysm clips, cardiac pacemakers, defibrillators, neurostimulators, cochlear implants, spinal cord stimulators, insulin or infusion pumps, metallic prostheses or fragments, heart valves, vascular stents, or shunts. surgical staples, clips, or joint replacements, radiation seeds, medication patches containing metal, or any other metallic or electronic implants)
* History of metallic injury to the eyes or body, or those with tattoos containing metallic ink, permanent makeup, or body piercings that cannot be removed.
* Any condition that poses a safety risk or could interfere with MRI scanning (e.g. severe claustrophobia or motion disorders or breathing problems, etc)

Psychiatric:

•History of hallucinogen persisting perception disorder (HPPD) (as per DSM-5 criteria)

Cardiovascular:

* Clinically significant cardiovascular conditions e.g., clinically significant EKG abnormalities, transient ischemic attack in the last 6 months, history of hemorrhagic stroke, history of myocardial infarction within 1 year of signing informed consent form (ICF)
* Baseline (heart rate < 60 bpm or > 90 bpm at screening or pre-dose
* Baseline hypertension (≥140 SBP or ≥90 DBP), after repeated measurements
* QTc Interval > 450msec on 12-lead EKG. Note: If QT-prolonging medications are started or increased in dose after enrollment and prior to dosing visit, a repeat EKG must be done >12-hours after this change to assure continued safe enrollment in the trial
* Clinically significant arrhythmia (e.g., uncontrolled atrial fibrillation, or untreated supraventricular tachycardia)
* Any current condition where physical activity is associated with palpitations, anginal pain or syncope

General health:

* Major systemic disorders, including seizure, insulin dependent diabetes mellitus, recent history (last 12 months) of advanced cancer or its treatment (radiation therapy or chemotherapy), had major surgery within 6 months from screening or plans to have surgery while enrolled in the study
* Inadequate hepatic function as determined by total bilirubin or alkaline phosphatase >3x institutional upper limit of normal; or aspartate aminotransferase (AST) or alanine transaminase (ALT) >3x institutional upper limit of normal. However, participants with Gilbert syndrome are allowed to enroll
* Inadequate renal function as determined by estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 (based on the MDRD equation)
* Participant is at increased risk of falls

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Acute changes in EEG-based ESBA | Pre- to post-dose two hours later
  Compare acute changes in EEG-based Lempel Ziv complexity (pre- to post-dose, arbitrary unit) between the four study arms, with the presence of biomarkers of AD pathology used in the statistical analyses as a moderator. Lempel-Ziv complexity in EEG is a non-linear analysis tool that quantifies the amount of entropy of spontaneous brain activity (ESBA).

SECONDARY OUTCOMES:
Changes in TNF-alpha | Screening to three weeks post dosing
  Compare changes in a biomarkers of neuroinflammation (TNF-alpha) psilocybin across the four study arms, with the presence of biomarkers of AD pathology used in the statistical analyses as a moderator. Reference Range 0.56-1.40 pg/mL

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Francisco, Sandler Neuroscience Building, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No